CLINICAL TRIAL: NCT04578847
Title: Prospective Non-randomized Stratified Study of REduction And DIscontinuation Treatment of TKI (Imatinib, Nilotinib, Dasatinib and Bosutinib) in Adults With Ph+ Chronic Myeloid Leukemia With Stable Deep Molecular Response
Brief Title: A Study of REduction And DIscontinuation Treatment of TKI (Imatinib, Nilotinib, Dasatinib and Bosutinib)
Acronym: READIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: READIT-2020
Record Dates: First submitted 2020-03-05; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Chronic Myeloid Leukemia; Chronic Myeloid Leukemia in Remission; BCR-ABL Positive Chronic Myelogenous Leukemia
Keywords: chronic myeloid leukimea; tyrosine kinase inhibitors; the TKI dose reduction; discontinuation treatment TKI; imatinib; nilotinib; dasatinib; bosutinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; nilotinib; Dasatinib; bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The TKI dose reduction (Experimental): Imatinib, nilotinib, dasatinib or bosutinib; the two stage of TKI dose reduction phase for 12 months (6 months and 6 months, respectively).
  Interventions: Drug: Imatinib; Drug: Nilotinib; Drug: Dasatinib; Drug: Bosutinib

INTERVENTIONS:
Drug: Imatinib — Initial dose - 400 mg daily. If on imatinib, the dose should be decreased to 300 mg daily on the first stage, to 200 mg daily - on the second stage.
Drug: Nilotinib — Initial dose - 300 or 400 mg twice daily. If on nilotinib to 400mg daily on the first stage, to 200 mg daily - on the second stage.
Drug: Dasatinib — Initial dose 100 or 140 mg daily. If on dasatinib then to 50 mg daily on the first stage, to 25 mg daily - on the second stage.
Drug: Bosutinib — Initial dose 500 mg daily. If on bosutinib, the dose should be reduced to 300 mg daily on the first stage, to 200 mg daily on the second stage.

SUMMARY:
The main goal of this study is to evaluate the stability of molecular response (major and deep molecular response( MMR and DMR)) in patients with chronic myeloid leukemia (CML) with stable DMR after two-stage dose reduction phase and discontinuation treatment TKI: imatinib, nilotinib, dasatinib and bosutinib.

DETAILED DESCRIPTION:
The duration of the dose reduction phase will be 12 months. This phase will have two stage of 6 months, respectively.

The dose of imatinib, nilotinib, dasatinib or bosutinib will be reduced by 25-50% on the first stage, and by another 25% on the second stage.

* The initial dose of imatinib will be 400 mg daily. The dose will be reduced by 300 mg daily on the first stage, by 200 mg daily - on the second stage.
* The initial dose of nilotinib will be 300 or 400 mg twice daily. The dose will be reduced by 400 mg daily on the first stage, by 200 mg daily - on the second stage.
* The initial dose of dasatinib will be 100 or 140 mg daily. The dose will be reduced by 50 mg daily on the first stage, by 25 mg daily - on the second stage.
* The initial dose of bosutinib will be 500 mg daily. The dose will be reduced by 300 mg daily on the first stage, by 200 mg daily - on the second stage.

All patients with stable deep molecular response (at least 2 years) will be included in treatment free remission phase (TFR-phase). The duration of TFR-phase will be 24 months.

The CML patients can enter the study already on reduced doses TKI, if they will meet the inclusion criteria.

It is possible to include patients, who have already received therapy with reduced doses of TKI. The duration of TKI therapy with reduced doses of 1 stage should be at least 6 months, if TKI doses meet of stage 1. The duration of TKI therapy with reduced doses of 2 stage should be for at least 6 months and the general duration of TKI therapy with reduced doses should be for at least 12 months, if TKI doses meet of stage 2.

ELIGIBILITY:
Inclusion Criteria:

1. CML in chronic phase.
2. TKI treatment for at least 3 years.
3. DMR (BCR-ABL≤0.01%) for at least 1 year, MMR (BCR-ABL≤0.1%) for at least 2 years
4. At least 3 molecular results over the preceding 24 months, which confirm the presence of MMR and DMR
5. Written Informed Consent
6. CML patients with DMR for at least 1 years and MMR for at least 2 years after STOP TKI in anamnesis.

For patients who are on the reduced dose TKI (1 stage) at the time of inclusion in the study

1. The duration of therapy at reduced doses of TKI phase I is at least 6 months.

For patients on the reduced dose TKI (2 stage, before TFR phase) at the time of inclusion in the study

1. DMR (BCR-ABL≤0.01%) for at least 2 years
2. The duration of therapy at reduced doses of TKI phase 1 is for at least 6 months, the total duration of therapy at reduced doses is for at least 12 months.

Exclusion Criteria:

1. Age under 18
2. ECOG >2
3. CML in accelerated phase or blast crisis at any time
4. Lack of Written Informed Consent
5. Pregnant or lactating women
6. Incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival, survival without molecular relapse | 37 months

SECONDARY OUTCOMES:
The proportion of patients with molecular relapse who achieved MMR and DMR after the resumption TKI therapy in standard doses | 37 months
The proportion of patients who resolved the adverse events after TKI dose reduction and discontinuation of TKI therapy | 37 months
The proportion of patients who have TKI withdrawal syndrome after TKI dose reduction and discontinuation of TKI therapy. | 37 months
Clinical factors, that affect the preservation of MMR after TKI dose reduction and discontinuation of therapy TKI. | 37 months
  sex (male, female)
Clinical factor, that affect the preservation of MMR after TKI dose reduction and discontinuation of therapy TKI. | 37 months
  age
Clinical factor, that affect the preservation of MMR after TKI dose reduction and discontinuation of therapy TKI. | 37 months
  risk group (Sokal, ELTS) at the time of diagnosis
Clinical factor, that affect the preservation of MMR after TKI dose reduction and discontinuation of therapy TKI. | 37 months
  duration of previous TKI treatment
Biological factor, that affect the preservation of MMR after TKI dose reduction and discontinuation of therapy TKI. | 37 months
  Duration of molecular response
Biological factor, that affect the preservation of MMR after TKI dose reduction and discontinuation of therapy TKI. | 37 months
  Molecular response at the time of inclusion in the study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Turkina, Professor, Principal Investigator — National Research Center for Hematology
Locations (1):
- National Research Center for Hematology, Moscow, Russia